CLINICAL TRIAL: NCT07284199
Title: A Multicenter Randomized Controlled Trial of the CA330 Haemoadsorption Device in Patients for Limiting Excess Anticoagulation in Non-elective caRdiac Surgery With Cardiopulmonary Bypass
Brief Title: CLEAR Trial: CA330 Cytokine Adsorption Column for Anticoagulant/Antiplatelet Patients in Non-Elective CPB Surgery.
Acronym: CLEAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Wuhan Asia Heart Hospital (Other); Xijing Hospital (Other); West China Hospital (Other); Guangdong Provincial People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Henan Provincial Chest Hospital (Other); Army Medical University, China (Other); Tongji Hospital (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-08-CLEAR
Record Dates: First submitted 2025-09-26; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: CABG; Aortic Dissection; Valvular Heart Diseases
MeSH Terms: conditions — Aortic Dissection; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CA330 Group (Experimental): CA330 Cytokine Adsorption Column and Standard Cardiopulmonary Bypass Management
  Interventions: Device: CA330 Cytokine Adsorption Column
- non-CA330 Group (No Intervention): Standard Cardiopulmonary Bypass Management Alone

INTERVENTIONS:
Device: CA330 Cytokine Adsorption Column — CA330 Cytokine Adsorption Column (Experimental Arm):
  The CA330 cytokine adsorption column is a novel hemoperfusion device integrated into the cardiopulmonary bypass (CPB) circuit. During CPB, the column removes specific circulating substances, including inflammatory mediators and residual anticoagulant/antiplatelet drugs, via adsorption. Patients in this arm will undergo non-elective cardiac surgery with standard anesthesia, surgery, and perioperative management, with the addition of the CA330 device placed inline during CPB.
  Arms: CA330 Group

SUMMARY:
The goal of this clinical trial is to evaluate whether the CA330 cytokine adsorption column can reduce perioperative severe bleeding adverse events in patients receiving anticoagulant and/or antiplatelet therapy who undergo non-elective cardiac surgery with cardiopulmonary bypass.

The main questions it aims to answer are:

* Does the use of the CA330 cytokine adsorption column lower the incidence of perioperative severe bleeding compared with standard care?
* Does the intervention improve short-term clinical outcomes, such as transfusion requirements, reoperation rates for bleeding, or overall postoperative recovery?

If there is a comparison group: Researchers will compare patients treated with the CA330 cytokine adsorption column versus patients receiving standard cardiopulmonary bypass management to see if cytokine adsorption provides additional safety and efficacy benefits.

Participants will:

* Undergo non-elective cardiac surgery requiring cardiopulmonary bypass.
* Be randomly assigned to receive either the CA330 cytokine adsorption column integrated into the CPB circuit (intervention arm) or standard CPB management without the device (control arm).
* Be monitored for perioperative bleeding outcomes, transfusion needs, reoperation rates, and overall postoperative prognosis.

DETAILED DESCRIPTION:
I. Study Background

Anticoagulant and antiplatelet agents reduce the risk of thrombosis by inhibiting platelet aggregation or coagulation factor activity, but they significantly increase the risk of intraoperative and postoperative bleeding. In urgent or emergency surgery, patients may be unable to discontinue anticoagulant or antiplatelet therapy in time, leading to markedly higher rates of bleeding complications during and after surgery. This presents major challenges for perioperative management and seriously affects patient outcomes.

The CA330 cytokine adsorption column is a novel hemoperfusion device that removes specific substances from the blood via adsorption during cardiopulmonary bypass (CPB). This study aims to evaluate the efficacy of CA330 in reducing perioperative severe bleeding adverse events during non-elective cardiac surgery under CPB in patients receiving anticoagulant or antiplatelet therapy. The ultimate goal is to provide a safer and more effective surgical strategy, improve patient prognosis, and generate high-level evidence for clinical practice.

II. Study Objectives

1. Primary Objective:

   To evaluate the efficacy of CA330 in reducing perioperative severe bleeding adverse events during non-elective cardiac surgery with CPB in patients receiving anticoagulant or antiplatelet therapy, thereby providing a safer and more effective surgical strategy.
2. Secondary Objectives:

By comparing perioperative outcomes and drug concentration monitoring between the intervention and control groups, to clarify the clearance efficiency of CA330 for different drugs during non-elective cardiac surgery with CPB, and to provide valuable guidance for clinical practice.

III. Study Protocol

1. Enrollment and Randomization:

   Eligible patients will be enrolled, randomized 1:1 into the intervention and control groups, provide written informed consent, and have baseline preoperative data collected.
2. Intervention and Procedures:

   * Standard anesthesia and surgical procedures will be applied.
   * CPB will be established using standardized management protocols based on guidelines and expert consensus.
   * In the intervention group, CA330 will be integrated into the CPB circuit; the control group will receive standard CPB management without the device.
   * Drug concentrations will be measured at:
   * T0: end of anesthesia induction
   * T1: initiation of CPB
   * T2: 30 min after CPB
   * T3: 60 min after CPB
   * T4: 120 min after CPB
   * T5: before weaning from CPB
   * T6: after protamine administration
   * Coagulation profile (five-item coagulation test) will be measured preoperatively and within 24h post-ICU admission.
   * Blood gas analysis will be performed at T0, T2, T5, and T6.
3. Outcome Measures:

   * Primary Endpoint:

   Incidence of BARC (Bleeding Academic Research Consortium) type 4 bleeding.
   * Secondary Endpoints:
   * Perioperative transfusion rate and volume of allogeneic blood products
   * Duration of mechanical ventilation
   * ICU length of stay
   * Total hospital length of stay
   * Hospital costs
   * Incidence of severe perioperative complications, including acute renal failure, severe hepatic dysfunction, myocardial infarction, ischemic stroke, and thromboembolic events.
4. Statistical Analysis:

   Comparative analyses will be performed between groups to assess differences in perioperative and follow-up outcomes, thereby determining the safety and efficacy of CA330 in non-elective cardiac surgery with CPB among patients receiving anticoagulant or antiplatelet therapy, and to guide optimal clinical management.
5. Sample Size:

A total of 120 patients are planned for enrollment. After enrollment of the first 60 patients, an interim analysis will be conducted based on observed endpoint outcomes to re-estimate sample size. The final sample size will not exceed 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo non-elective cardiovascular surgery requiring cardiopulmonary bypass;
* Patients currently receiving one or more of the following medications - indobufen, ticagrelor, warfarin, cilostazol, dabigatran, rivaroxaban, or apixaban - with the last dose administered within the drug washout period.

Exclusion Criteria:

* Patients with a history of chronic liver failure, stage 5 chronic kidney disease (CKD5), or requiring regular dialysis;
* Patients in special physiological states: pregnancy or puerperium;
* Patients with advanced-stage malignancy or scheduled cardiovascular surgery related to tumor management;
* Patients with allergic reactions to cytokine adsorption column resin or related components;
* Patients with known bleeding risk due to hematologic disorders such as heparin-induced thrombocytopenia, hemophilia, or acute sickle cell crisis;
* Patients with severe infection, including severe sepsis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of BARC-4 severe bleeding | within 48 hours of the perioperative period
  The primary endpoint is a composite outcome, defined as the occurrence of any one of the following events:
  1. Intracranial hemorrhage within 48 hours of the perioperative period(Number);
  2. Reoperation after sternotomy closure to control bleeding(Number);
  3. Transfusion of ≥5 units (1,000 mL) of whole blood or packed red blood cells within 48 hours(Number);
  4. Postoperative chest drainage ≥2 L within 24 hours(Number).
  Unit of measure: number of participants experiencing at least one component of the composite endpoint.

SECONDARY OUTCOMES:
All-cause mortality(Death from any cause). | From the end of surgery to 30 days postoperatively
  Unit of Measure: Number (%)
Volume and incidence of perioperative allogeneic blood product transfusion | From the end of surgery to 30 days postoperatively
  Unit of Measure: Number (%)
Total Volume of Allogeneic Blood Products Transfused | From the end of surgery to 30 days postoperatively
  Unit of Measure: mL
Incidence of other severe complications, including new-onset perioperative renal failure, severe hepatic dysfunction, myocardial infarction, ischemic stroke, and thromboembolic events | From the end of surgery to 30 days postoperatively
  Unit of Measure: Number (%)
ICU length of stay | From the end of surgery to 30 days postoperatively
  Unit of Measure: Days
Hospital length of stay | From the end of surgery to 30 days postoperatively
  Unit of Measure: Days
Hospitalization costs | From the end of surgery to 30 days postoperatively
  Unit of Measure: CNY

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Hou, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Center for Cardiac Intensive Care, Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China